CLINICAL TRIAL: NCT02095197
Title: A Prospective Randomized Controlled Trial of Standardized C7-T1 Epidural Steroid Injections Versus Targeted Injection Via Cervical Epidural Catheter for the Treatment of Cervical Radicular Pain
Brief Title: C7-T1 Epidural Steroid Injections Versus Targeted Injection for Treatment of Cervical Radicular Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Associate Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00089080; STU00089080 (Other: Northwestern University IRB)
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Radicular; Neuropathic, Cervical; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Catheter delivery (Other): Cervical epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
  No Catheter Delivery will be used to deliver the medication.
  Interventions: Drug: Triamcinolone 80mg
- Catheter targeted delivery (Active Comparator): Cervical epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
  Catheter targeted delivery will be used to deliver the medication.
  Interventions: Drug: Triamcinolone 80mg

INTERVENTIONS:
Drug: Triamcinolone 80mg — C7-T1 Cervical interlaminar epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
  Other Names: Kenalog

SUMMARY:
Cervical radicular pain is a common, disabling problem, occurs in 83:100,000 individuals per year. Symptoms are most often caused by intervertebral disc herniation (21.9%) or central or foraminal stenosis from spondylosis (68.4%). Patients complain of pain in the head, neck, scapula or arm. The diagnosis of radicular pain is made clinically by history and physical examination, supported by imaging studies and electrodiagnostic tests. No study has compared the differences in pain, medication utilization, functional outcomes, or patient satisfaction between interlaminar and targeted epidural injections in the cervical spine. In theory, the technique of targeted epidural steroid delivery with a catheter has a lower risk of accidental vascular trespass or disc penetration during the procedure, and far less risk of dural penetration or spinal cord injury at rostral levels of the cervical spinal cord as compared with the interlaminar technique. The investigators hypothesize that this technique results in superior pain control, decreased medication use, improved function and fewer repeat injections. This data could improve patient safety and affect the evolving treatment guidelines for cervical epidural injections.

DETAILED DESCRIPTION:
Cervical radicular pain is a common, painful, disabling problem, often treated by epidural steroid injection (ESI). Two techniques of steroid delivery into the cervical epidural space include the transforaminal and interlaminar approaches. We aimed to determine if the CIESI with versus without a catheter is associated with superior clinical outcomes at follow-up. We hypothesized that the use of a targeted epidural catheter technique would result in superior pain control, function, decreased analgesic use, and lower surgical incidence as compared to standard CIESI at C7-T1.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 18-75 with C2-6 unilateral radicular pain who are scheduled to undergo cervical epidural steroid injection treatment.
* Pain lasting greater than 2 weeks.
* Pain resistant to a trial of conservative therapy (i.e. oral steroids,nonsteroidal anti-inflammatory drugs, opioids, muscle relaxants, physical therapy or chiropractic care)

Exclusion Criteria:

* Patient refusal.
* Lack of consent.
* Systemic infection or local infection over planned injection site in posterior cervical spine.
* Bleeding disorder, current use of anticoagulants or anti-platelet medications.
* Intrinsic spinal cord lesions in the cervical region.
* History of central neurologic, cerebrovascular, demyelinating or muscular disease.
* Concomitant use of oral or injected steroids.
* Allergy to medications being used for injection procedures.
* Inability to communicate with staff or to participate in follow up.
* Pregnancy.
* Inability to perform handgrip or arm strength testing.
* Cognitive deficit or motor neuron disease.
* Daily opiate use that preceded the onset of cervical radicular symptoms or daily opiate use exceeding 3 months prior to study inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Walega, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCormick ZL, Nelson A, Bhave M, Zhukalin M, Kendall M, McCarthy RJ, Khan D, Nagpal G, Walega DR. A Prospective Randomized Comparative Trial of Targeted Steroid Injection Via Epidural Catheter Versus Standard C7-T1 Interlaminar Approach for the Treatment of Unilateral Cervical Radicular Pain. Reg Anesth Pain Med. 2017 Jan-Feb;42(1):82-89. doi: 10.1097/AAP.0000000000000521. PMID 27922950

RESULTS

PARTICIPANT FLOW:
Groups:
- No Catheter Delivery: Cervical epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
  No Catheter Delivery will be used to deliver the medication.
  Triamcinolone 80mg: C7-T1 Cervical interlaminar epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
- Catheter Targeted Delivery: Cervical epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
  Catheter targeted delivery will be used to deliver the medication.
  Triamcinolone 80mg: C7-T1 Cervical interlaminar epidural steroid injection with Triamcinolone 80mg and 1 mL 1% lidocaine. Total volume is 2 cc.
Period: Overall Study
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery
Started | 40 | 39
Completed | 40 | 36
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery | Total
Number analyzed (Participants) | 40 | 36 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 32 | 69
  >=65 years | 3 | 4 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [39 to 56] | 50 [45 to 60] | 49 [42 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 40 | 36 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥50% Pain Reduction on the Numeric Rating Score (NRS) for Pain
Description: The percentage of participants who reported ≥50% pain reduction on the numeric rating score for pain at the 1 month follow-up assessment period.
  Numeric Rating Scale (NRS) for pain consists of a range where 0 (is no pain) and 10 (is extreme pain).
  Percentage of participants with pain reduction = 100% (number of participants with pain reduction/all participants)
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery
Number analyzed (Participants) | 38 | 36
percentage of participants | 60 [45 to 75] | 72 [57 to 87]
Statistical Analysis 1: Comparison: No Catheter Delivery vs Catheter Targeted Delivery; Test type: Superiority or Other; p = 0.23, Fisher Exact

2. Secondary Outcome: Decrease of > 6.8 Point Reduction in Medication Quntification Scale (MQS-III)
Description: The Medication Quantification Scale was designed as a method of quantifying different drug regimens (Harden et al, Journal of Pain, 2005). The detriment weights derived from the healthcare survey for each of the 22 medication classes are the critical values that when multiplied by a dosage score it gives a patient MQS score. It computes a single numeric value for a patient's pain medication profile. We recorded the names and doses of each medication being used then quantified the total burden of each subject's medication using the MQS-III. which assigns a measurement to each drug based on both the dose taken and its burdensomeness (derived from expert consensus).
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery
Number analyzed (Participants) | 40 | 36
Participants | 13 | 9
Statistical Analysis 1: Comparison: No Catheter Delivery vs Catheter Targeted Delivery; Test type: Superiority or Other; p = 0.47, Chi-squared

3. Secondary Outcome: Patient Global Impression of Change Score (PGIC) Less Than 3
Description: PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as:
  1=Very Much Improved, 2=Much Improved, 3=Minimally Improved, 4=No Change, 5=Minimally Worse, 6=Much Worse, 7=Very Much Worse.
  A PGIC score less than 3 means the patient reported "much improved" to "very much improved."
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery
Number analyzed (Participants) | 40 | 36
Participants | 22 | 24
Statistical Analysis 1: Comparison: No Catheter Delivery vs Catheter Targeted Delivery; Test type: Superiority or Other; p = 0.30, Chi-squared

4. Secondary Outcome: Greater Than or Equal to a 30% Reduction in Oswestry Neck Disability Index Score
Description: This questionnaire has been designed to give us information to how neck pain has affected the ability to manage in everyday life. There are ten sections, 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. All the points can be summed to a total score. The maximum points scored is 50. The reported score divided by 50 is then transformed to a percentage score by multiplying by 100. The Minimum dectectable change (90 % confidence) is 5 points or 10 percent.
Time Frame: 1 month
Population: Both demonstrate a difference from pretreatment baseline (P=0.05).
Measure: Count of Participants; unit: Participants
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery
Number analyzed (Participants) | 40 | 36
Participants | 23 | 24
Statistical Analysis 1: Comparison: No Catheter Delivery vs Catheter Targeted Delivery; Test type: Superiority or Other; p = 0.41, Chi-squared

ADVERSE EVENTS:
Arm/Group | No Catheter Delivery | Catheter Targeted Delivery
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/36
Other Adverse Events (participants affected / at risk) | 0/40 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes